CLINICAL TRIAL: NCT02793089
Title: Retrospective Cohort Study of Increased Risk of Ectopic Pregnancy Associated With Marked Variation of Estradiol During the Early Luteal Phase and High Progesterone on hCG Day in IVF
Brief Title: Risk of Ectopic Pregnancy and Variation of Luteal Estradiol and Progesterone Levels in IVF
Status: Completed | Type: Observational
Sponsor: IVI Vigo (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1409-VGO-059-EM
Record Dates: First submitted 2016-05-18; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- First quartile: No drugs are administered. It is an observational study. Collect retrospectively data.Analysis of Ectopic Pregnancy incidence through Estradiol (E2) and progesterone (P4) levels on hCG day and seven days later (hCG+7).
  Interventions: Other: Analysis of Ectopic Pregnancy incidence
- Second quartile: No drugs are administered. It is an observational study. Collect retrospectively data.Analysis of Ectopic Pregnancy incidence through Estradiol (E2) and progesterone (P4) levels on hCG day and seven days later (hCG+7).
  Interventions: Other: Analysis of Ectopic Pregnancy incidence
- Third quartile: No drugs are administered. It is an observational study. Collect retrospectively data.Analysis of Ectopic Pregnancy incidence through Estradiol (E2) and progesterone (P4) levels on hCG day and seven days later (hCG+7)
  Interventions: Other: Analysis of Ectopic Pregnancy incidence
- Fourth quartile: No drugs are administered. It is an observational study. Collect retrospectively data.Analysis of Ectopic Pregnancy incidence through Estradiol (E2) and progesterone (P4) levels on hCG day and seven days later (hCG+7)
  Interventions: Other: Analysis of Ectopic Pregnancy incidence

INTERVENTIONS:
Other: Analysis of Ectopic Pregnancy incidence — Collect retrospectively data. Analysis of Ectopic Pregnancy incidence through Estradiol (E2) and progesterone (P4) levels on hCG day and seven days later (hCG+7)

SUMMARY:
This study evaluates the increased risk of ectopic pregnancy associated with marked variation of estradiol during the early luteal phase and high progesterone on hCG day in IVF.

DETAILED DESCRIPTION:
This is a retrospective cohort study of 578 patients who had no risk of EP (672 fresh transfer IVF cycles) between January 2005 and December 2014. Few studies have reported the relation between hormonal levels and ectopic pregnancy (EP) in IVF. Investigators describe EP incidence according to estradiol (E2) and progesterone (P4) levels on hCG day and seven days later (hCG+7) or their variation between both days.

ELIGIBILITY:
Inclusion Criteria:

* Normal Fallopian tubes in HSG and /or laparoscopy
* Normal Uterus: Abscence of myomas and Müllerian anomalies .

Exclusion Criteria:

* Previous Ectopic Pregnancy .
* Recurrent Abortion .
* Tubal Factor : pelvic inflammatory disease, Hydrosalpinx
* Previous abdominal surgery (except laparoscopy) .
* Prior Peritonitis
* Smoking (at least 1 cigarette/day) .

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who had no risk of EP (672 fresh transfer IVF cycles) between January 2005 and December 2014.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2005-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Ectopic pregnancy rate | Up to 108 months

CONTACTS AND LOCATIONS:
Overall Officials: Elkin Muñoz, Principal Investigator — IVI Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosch E, Labarta E, Crespo J, Simon C, Remohi J, Jenkins J, Pellicer A. Circulating progesterone levels and ongoing pregnancy rates in controlled ovarian stimulation cycles for in vitro fertilization: analysis of over 4000 cycles. Hum Reprod. 2010 Aug;25(8):2092-100. doi: 10.1093/humrep/deq125. Epub 2010 Jun 10. PMID 20539042
- [Background] Paltieli Y, Eibschitz I, Ziskind G, Ohel G, Silbermann M, Weichselbaum A. High progesterone levels and ciliary dysfunction--a possible cause of ectopic pregnancy. J Assist Reprod Genet. 2000 Feb;17(2):103-6. doi: 10.1023/a:1009465900824. PMID 10806589
- [Result] Cobo A, Bosch E, Alvarez C, de los Santos MJ, Pellicer A, Remohi J. Effect of a sharp serum oestradiol fall before HCG administration during ovarian stimulation in donors. Reprod Biomed Online. 2007 Aug;15(2):169-74. doi: 10.1016/s1472-6483(10)60705-5. PMID 17697492